CLINICAL TRIAL: NCT05350111
Title: CArdioMetabolic Prevention in Adolescents With Body Weight Issues: the Effect of Group Intervention and Telemedicine
Brief Title: CArdioMetabolic Prevention in Adolescents
Acronym: CAMP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Faculty Hospital Kralovske Vinohrady (Other Government)
Responsible Party: Principal Investigator, Irena Aldhoon Hainerova, Assoc. Prof. M.D., Ph.D., Faculty Hospital Kralovske Vinohrady
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KDD FNKV
Record Dates: First submitted 2022-03-29; First posted 2022-04-27 (Actual); Last update posted 2022-04-27 (Actual); Status verified 2022-04

CONDITIONS: Adolescent Obesity; Life Style, Healthy; Body Weight Changes; Cardiometabolic Syndrome
Keywords: adolescents; obesity; cardiometabolic health; telemedicine
MeSH Terms: conditions — Pediatric Obesity; Body Weight Changes; Metabolic Syndrome; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- group supported through group education and telemedicine tools (Other): the group of this pilot study will be compared to conventional obesity clinic
  Interventions: Behavioral: lifestyle education

INTERVENTIONS:
Behavioral: lifestyle education — education on healthy lifestyle through group sessions and telemedicine tools

SUMMARY:
The aim of the CArdioMetabolic Prevention (CAMP) pilot study is to investigate the effect of a group intervention on lifestyle in adolescents and on at least one adult family member. This will be followed by telemedicine tools for 12-week-time period. A face-to-face group intervention addressing nutrition, physical activity and well being together with an assessment of anthropometry parameters, body composition, questionnaires, blood and stool sampling will be done before and after 12 weeks of telemedicine.

The study aims to investigate:

* the effect of 12-week intervention on body weight, anthropometry parameters and cardiometabolic markers in comparison to the conventionally led obesity clinic for adolescents
* the compliance with telemedicine tools that will focus on the support of balance nutrition, physical activity (evaluation of daily steps through smart bands) and family well being in regards to the effect on anthropometry and laboratory parameters
* the effect of the intervention on data from questionnaires (eating disorders, quality of life, psychological health) before and after the intervention
* data analysis of family members with respect to theirs offspring

DETAILED DESCRIPTION:
In a 12-month pilot study it is expected to include four groups composed of 10-12 adolescent participants with increased body weight. The participants will be recruited from new patients attending pediatric endocrine clinics in the Department of Children and Adolescents of Faculty Hospital Kralovske Vinohrady and Third Faculty of Medicine Charles University.

For those included, a detailed history, laboratory (routine investigation additionally to serum storage and stool for microbiome analysis) and physical examination will be assessed during the initial visit in the outpatient clinic. During one day group intervention each adolescent with at least one family member will undergo education session on nutrition, healthy eating and physiological support incl. cognitive behavioral sessions. There will be an assessment of individual fitness and participants will try different suitable options to increase their daily physical activity. Participants will be asked to bring filled questionnaires that address different aspects of lifestyle and psychological well being. A detailed anthropometry examination and body composition will also be performed. An ultrasound examination of carotid intima-media thickness and visceral fat mass measurements will be assessed in all adolescents. The body composition, body weight and height will also be measured in all accompanied family members. All participants will receive smart bands for the following 12 weeks to support physical activity and monitor their daily step count.

This group intervention will be followed by a12-week time period in which telemedicine tools and frequent virtual contacts will be done to support family healthy lifestyle.

After 12 weeks a group session will be undertaken in order to evaluate all aspects of lifestyle through repeated questionnaire survey. Laboratory, ultrasound and anthropometry examination will be done in order to monitor the effect of this intervention and compared to participants visiting the conventional obesity clinic of our hospital. A further follow-up will be offered to all participants.

ELIGIBILITY:
Inclusion Criteria:

* age range: 12-19 years
* diagnosis of obesity = body mass index (in kg/m2) above 97th centile for age and sex
* obesity likely due to impaired healthy lifestyle

Exclusion Criteria

* genetic forms of obesity
* obesity due to endocrinopathy

Ages: 12 Years to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-03-27 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Effect on anthropometry parameters | 12 weeks
  change of z-score of body mass index (in kg/m2) before and after the 12-week intervention (successful intervention should lead to a decline of z-score BMI)
Effect on depression | 12 weeks
  change in Beck depression score before and after the 12 weeks of intervention (range: 0-60 points, no depression = 0-10 points, mild depression = 10-20 points, moderate depression = 20-40 points, severe depression = 40-60 points)
Effect on fitness | 12 weeks
  change of fitness level assessed by 6-minute walk test before and after the 12 weeks of intervention (evaluated by the distance reached within the 6-minute walk test)
Effect on quality of life | 12 weeks
  change of score of quality of life (assessed by KIDSCREEN questionnaire, the higher the score, the higher quality of life)
Effect on eating behavior | 12 weeks
  change of score assessing cognitive restraint (greater the score, greater the restraint), disinhibition of control over eating (greater the score, greater the disinhibition) and perceived hunger (greater the score, greater the hunger) via Eating Inventory questionnaire before and after the 12 weeks of intervention

SECONDARY OUTCOMES:
Effect on body composition of an accompanied adult person | 12 weeks
  change of percentage of fat mass assessed by bioimpedance before and after the 12-week intervention
Effect on body weight of an accompanied adult person | 12 weeks
  change of body weight in kg before and after the 12-week intervention

CONTACTS AND LOCATIONS:
Overall Officials: Irena D Aldhoon Hainerova, MD PhD, Principal Investigator — Fakultní nemocnice Královské Vinohrady
Locations (1):
- Faculty Hospital Kralovske Vinohrady, Prague, Czechia